CLINICAL TRIAL: NCT05198583
Title: Executive Function and Brain Development in Adolescents With Severe Congenital Heart Disease (Teen Heart Study)
Brief Title: EF Intervention in Children With Severe Congenital Heart Disease
Acronym: E-FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Teen Heart Intervention
Record Dates: First submitted 2021-12-07; First posted 2022-01-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Heart Defects, Congenital; Executive Dysfunction
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will have a play-based intervention, including online games, analogue card games as well as a weekly coaching session to enhance executive functions.
  Interventions: Other: E-Fit
- Control (No Intervention): The control group will get access to the online games, a list of the analogue card games used and fact sheets about possibilities to enhance executive functions in everyday life (which are used in the intervention group during the coachings) after finishing the study.

INTERVENTIONS:
Other: E-Fit — The intervention lasts a total of 8 weeks and is structured in 3 modules. The first module consists of a weekly strategy training in which problems resulting from executive dysfunction are addressed. Online games form the second module. These are games implemented online to promote EF through play. The third module is also based on games: The families receive several board games to play together at home. This third module is voluntary.
  Arms: Intervention

SUMMARY:
Survival rates of children with severe congenital heart disease (CHD) have increased with ongoing medical progress over the past decades. However, many children with CHD face academic challenges during adolescence, which are associated with executive dysfunction. Executive functions (EF), higher-order cognitive processes allowing goal-directed behavior, can be particularly affected in children with CHD. To improve EF in affected children, a specific EF intervention has been developed.

The intervention lasts a total of 8 weeks and is structured in 3 modules. The first module consists of a weekly strategy training in which problems resulting from executive dysfunction are addressed. Online games form the second module. These are games implemented online to promote EF through play. The third module is also based on games: The families receive several board games to play together at home. This third module is voluntary. This intervention is tested on its feasibility. As the intervention was built in a patient centered manner, we expect it to be feasible, showing in a high adherence rate and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Born with CHD
* Underwent cardiopulmonary bypass surgery
* No genetic syndrome detected, no known dysmorphic-syndrome
* Aged 10 to 12
* written informed consent of parents and verbal informed consent of children
* EF deficits showing in screening

Exclusion Criteria:

* Failure to provide a signed Informed Consent
* Heart surgery without cardiopulmonary bypass
* Heart surgery not performed in Switzerland
* Any genetic syndrome detected
* large cerebral lesions (stroke, HIE) or severely neurologically impaired as a result of a serious event

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Fun and cognitive demand | 5 minutes
  Subjective Feasibility, Fun and cognitive demand:
  the two questions "How fun was the training?" and "How much did you use your brain" are answered on a 5-point Likert scale (1 referring to not at all and 5 referring to very much). Both questions are treated as ordinal scaled and median and interquartile range will be reported.
Children's Feeling Scale | 5 minutes
  Subjective Feasibility, Affect 11-point single item bipolar scale (-5 referring to "very bad" and 5 referring to "very good"). The Hulley feeling scale is treated as ordinal scaled and median and interquartile range will be reported.
Acceptance and Feasibility scale | 5 minutes
  4-point Likert scale (1 referring to "don't agree at all" and 4 referring to "fully agree"). Treated as ordinal scaled and median and interquartile range, as well as percentages of persons who answered the items with 3 or 4, will be reported.
Completion rate (Objective Feasibility): | 5 minutes
  Frequency (amount of participants who completed the training)/(total amount of participants enrolled)
Observed engagement | 2 minutes
  Engagement of the participant during coaching sessions rated on a 7-point Likert scale
Session data | 5 minutes
  duration, number of completed sessions, and for the computerized training, the coaching, and the card games
Recruitment rate | 5 minutes
  amount of participants who agreed to participate/amount of invited participants
E-Fit Fidelity Measurement System tool | 8 hours
  Tool to check whether the intervention was implemented as intended, answered by "yes" and "no" for each item
Feedback in coaching sessions | 5 minutes
  qualitative feedback during the sessions about practicality of the intervention
Observed involvement | 5 minutes
  involvement of the coach rated in 3 questions on a 7-point Likert scale
Session rating scale | 2 minutes
  4 questions about the practicality of the session rated by the participant
Retention rate | 2 minutes
  participants who finished the study/participants who enrolled
Occurrence of adverse events (AEs) | From Start of the study until the end of the study, assessed up to 25 months
  Amount of adverse events
Behavior Rating Inventory of Executive Function (BRIEF) | 15 minutes
  The BRIEF assesses Executive Functions Behavior in everyday life. The results will be be transformed into a categorical variable with results > 1 SD defined as abnormal (T-scale >= 60).
Color word Interference Task (D-KEFS) | 5 minutes
  The D-KEFS Color-Word Interference Test is based on the classic Stroop task, which is primarily used to assess the ability to inhibit verbal responses (inhibition).
Go/NoGo Test battery for attention testing (TAP) | 5 minutes
  In this test, 2 implementation forms with different stimulus material are offered. In the 1st condition, reaction times and errors are measured in a simple "Go/Nogo" condition with two stimuli (+ and x: 2 stimuli, one critical), in the 2nd more complex condition with 5 squares with different filling patterns, 2 of which are defined as critical (5 stimuli, 2 critical).
Trail-Making-Test (D-KEFS) | 5 minutes
  The D-KEFS Trail Making Test is a revision and extension of the classic alternating number and letter matching task, which is known as a proven instrument for assessing cognitive flexibility. With the help of four additional conditions, the basic abilities of visual scanning, connecting numbers and letters, and motor speed can be assessed. This results in a differentiated overall picture of the interaction of different basic and higher cognitive abilities.
Number-Letter-sequencing (WISC-V) | 10 minutes
  In number repeating, the subject is read a sequence of numbers and asked to repeat them in the same order (number repeating - forwards), in reverse order (number repeating - backwards) or in ascending order (number repeating - sequential).
Tower Task from the (D-KEFS) | 15 minutes
  The D-KEFS Tower Test is a revision of classic tower tasks in which discs are to be restacked with the help of three rods in such a way that given tower templates are replicated, while observing certain rules. Nine standardised tasks covering a difficulty spectrum from very easy to very difficult are designed to avoid floor and ceiling effects. The test measures, among other things, spatial planning ability, rule learning, inhibition of impulsive or perseverative response behaviour, as well as the development and maintenance of mental attitudes.
Balloon Analogue Risk Task (BART) | 10 minutes
  In the experiment, participants are presented with a balloon. The participant is prompted to inflate the balloon using the Right Arrow key. After successfully inflating the balloon by 1 unit, the participant receives five points. The more the participant inflates the balloon, the more points they receive. E-Prime randomly selects a number between 1 and 100 for each trial representing the total number of inflated units before the balloon bursts. If the participant inflates the balloon too much, it pops and no points are given. Participants also have the choice to press the Left Arrow to advance the trial while keeping their points. There is one practice trial and 5 critical trials.

SECONDARY OUTCOMES:
The Family Relationship Index | 10 minutes
  27 questions answered "does apply" or "does not apply"
Kidscreen-10 | 5 minutes
  10 questions to assess the child's subjective health and well-being on a 5-point Likert scale
Kidscreen-27 | 10-15 minutes
  27 questions to assess the child's health and well-being from a parent's perspective on a 5-point Likert scale
short form of the Conners-3 | 20 minutes
  42 questions answered on a 4-point Likert scale and 2 open questions to screen for behavioral problems
Social Responsiveness Scale | 20 minutes
  65 questions answered on a 4-point Likert scale to screen for behavioral problems
Resilience Scale | 5 minutes
  13 questions answered on a 7-point Likert scale to assess resilience by acceptance of self-, life- and personal competencies

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Schmid AS, Ehrler M, Wehrle F, Tuura RO, Kretschmar O, Landolt M, Latal B. Multimodal personalised executive function intervention (E-Fit) for school-aged children with complex congenital heart disease: protocol for a randomised controlled feasibility study. BMJ Open. 2023 Nov 9;13(11):e073345. doi: 10.1136/bmjopen-2023-073345. PMID 37945305